CLINICAL TRIAL: NCT02125357
Title: A Randomized Phase II Study of Sequencing Abiraterone Acetate and Enzalutamide in Metastatic Castration-Resistant Prostate Cancer
Brief Title: Sequencing Abiraterone and Enzalutamide in mCRPC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GUTG-001
Record Dates: First submitted 2014-04-22; First posted 2014-04-29 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: sequencing; abiraterone; enzalutamide; metastatic castration-resistant prostate cancer; randomized
MeSH Terms: interventions — Abiraterone Acetate; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A - Abiraterone Acetate (Other): Abiraterone acetate 1000mg PO OD with prednisone 5mg PO BID or 10mg OD as per standard of care, or until PSA progression then cross-over to Arm B.
  Interventions: Drug: Abiraterone acetate
- B - Enzalutamide (Other): 160mg PO OD as per standard of care, or until PSA progression then cross-over to Arm A.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Abiraterone acetate — Abiraterone acetate 1000mg PO OD with prednisone 5mg PO BID or 10mg OD as per standard of care.
  Other Names: Zytiga
  Arms: A - Abiraterone Acetate
Drug: Enzalutamide — 160mg PO OD as per standard of care.
  Other Names: Xtandi
  Arms: B - Enzalutamide

SUMMARY:
This study is being offered to patients who have castrate-resistant (also known as hormone-refractory) prostate cancer. The cancer has metastasized or spread outside the prostate area to other parts of the body.

The purpose of this study is to evaluate the effects of sequencing hormonal therapies (abiraterone acetate and enzalutamide) and to assess treatment efficacy of these two agents.

DETAILED DESCRIPTION:
Abiraterone acetate and enzalutamide have emerged as standard therapies in metastatic castration-resistant prostate cancer (mCRPC). Both agents improve outcomes in patients previously treated with docetaxel and in those that are chemotherapy-naive. Although their mechanisms of action differ, both abiraterone and enzalutamide target persistent androgen receptor (AR) signaling. Abiraterone inhibits CYP17 and testicular and extragonadal androgen production whereas enzalutamide directly antagonises the AR. Whether cross resistance occurs between these agents if used in sequence is unknown, but theoretically disparate mechanisms of resistance may allow for successful sequencing of these agents. Prior studies have reported Prostate-Specific Antigen (PSA) response rates of under 10% in patients treated with abiraterone after enzalutamide and 13%-29% in patients treated with enzalutamide after abiraterone. Since these data were generated in small, retrospective series, a prospective clinical trial is warranted to evaluate effects of sequencing abiraterone and enzalutamide. A randomised phase II study is proposed in which patients with PSA progression on abiraterone or enzalutamide will be crossed over to the opposite agent. Although not a surrogate for clinical outcomes, PSA changes will be used to assess treatment efficacy since PSA expression is driven by AR activation.

Apart from determining optimal sequencing of abiraterone and enzalutamide in mCRPC patients, a key issue associated with the use of these agents is identifying circulating biomarkers associated with treatment response and resistance. Our group has preliminary data showing that a high proportion of enzalutamide-resistant mCRPC patients and some abiraterone-resistant mCRPC patients possess focal AR amplification in cell-free tumour DNA extracted from plasma. In pre-clinical studies, other potential mechanisms of resistance to these agents include increased expression of AR splice variants (abiraterone and enzalutamide) increased expression of CYP17 (abiraterone), upregulation of the stress-activated chaperone protein clusterin (enzalutamide only) and a point mutation (F876L) in the ligand-binding domain of the AR (enzalutamide only). Non-coding RNAs (ncRNAs) are additional biomarkers of interest since they are implicated in tumorigenesis and are readily detectable in plasma of mCRPC patients. Examination of these biomarkers in serum and plasma is planned, with the aim of identifying potentially novel factors associated with treatment efficacy and resistance in mCRPC patients receiving abiraterone and enzalutamide.

The cognitive effects of abiraterone and enzalutamide are not well described. Enzalutamide is known to cross the blood-brain barrier and infrequently causes seizures, possibly related to effects on the γ-aminobutyric acid-gated chloride channel. In the enzalutamide registration study, a small subset (< 5%) of patients also developed mental impairment disorders including amnesia, memory impairment, cognitive disorder and disturbance in attention. Conversely, no central nervous system effects of abiraterone have been reported. Cognitive testing will therefore be undertaken in this study to evaluate potential differences between these agents.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent
2. Adult males ≥ 18 years age
3. History of adenocarcinoma of the prostate diagnosed histologically without evidence of neuroendocrine or small cell differentiation
4. Prior surgical orchiectomy or if on luteinizing hormone-releasing hormone (LHRH) agonist/antagonist then testosterone < 1.7 nmol/L at screening visit (patients must maintain LHRH agonist/antagonist therapy for duration of study treatment if not surgically castrated)
5. Evidence of metastatic disease on bone scan or CT scan
6. Evidence of biochemical or imaging progression in the setting of surgical or medical castration. Progressive disease for study entry is defined by one of the following three criteria:

   1. PSA progression: minimum of two rising PSA values from a baseline measurement with an interval of ≥ 1 week between each measurement. Minimum PSA at screening visit is > 2.0 ug/L
   2. Soft tissue or visceral disease progression (see Appendix B for definition of measurable disease as per Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 criteria)
   3. Bone progression: ≥ 2 new lesions on bone scan
7. ECOG performance status 0-2 (see Appendix C)
8. Eligible for treatment with either abiraterone acetate or enzalutamide as per standard of care guidelines
9. Adequate organ function defined as:

   1. Absolute neutrophil count ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L and hemoglobin ≥ 80 g/L
   2. Creatinine clearance ≥ 30 ml/min (calculated by Cockcroft-Gault formula, see Appendix D)
   3. Serum potassium within normal limits
   4. Total bilirubin ≤ 1.5 x upper limit of normal (ULN) except for patients with known Gilbert's syndrome (direct bilirubin ≤ 1.5 x ULN)
   5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x ULN
10. Able to swallow study drug and comply with study requirements including provision of peripheral blood samples at specified time points for correlative studies
11. Recovery from all prior treatment-related toxicity to grade ≤ 2 (as per Common Terminology Criteria for Adverse Events 4.0)

Exclusion Criteria:

1. Severe concurrent illness or co-morbid disease that would make the subject unsuitable for enrolment
2. Prior therapy with CYP17 inhibitors (including abiraterone acetate, TAK-700, TOK-001 and ketoconazole), enzalutamide or other experimental anti-androgens (e.g. ARN-509, TOK-001)
3. Prior systemic chemotherapy for mCRPC
4. Life expectancy < 6 months
5. Active concurrent malignancy (with the exception of non-melanomatous skin cancer)
6. Wide-field radiotherapy or radioisotopes such as Strontium-89 or Radium-223 ≤ 28 days prior to starting study drug (limited-field palliative radiotherapy for 1-5 fractions is permitted at anytime prior to commencement protocol therapy)
7. Brain metastases or active epidural disease (treated epidural disease is permitted)
8. Use of herbal products that may lower PSA level (e.g. saw palmetto)
9. Contraindication to prednisone therapy including poorly controlled diabetes mellitus
10. History of seizure or seizure disorder, or history of any cerebrovascular event within 6 months of study entry.
11. Gastrointestinal disorder affecting absorption
12. Major surgery within 4 weeks of starting study treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
PSA response rate in mCRPC patients with PSA progression on first-line therapy when crossed over to second-line therapy with the opposite agent | 1 year

SECONDARY OUTCOMES:
Potential biomarkers that are associated with treatment efficacy and/ or resistance | 1 year
  Among mCRPC patients receiving abiraterone acetate and enzalutamide

OTHER OUTCOMES:
PSA response rate in mCRPC patients treated with first-line abiraterone acetate or enzalutamide | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kim N Chi, MD, Study Chair — British Columbia Cancer Agency
Locations (7):
- Canada (7):
  - BC Cancer Agency - Abbotsford, Abbotsford, British Columbia
  - BC Cancer Agency - Southern Interior, Kelowna, British Columbia
  - BC Cancer Agency - Centre for the North, Prince George, British Columbia
  - BC Cancer Agency - Fraser Valley, Surrey, British Columbia
  - Vancouver Prostate Centre, Vancouver, British Columbia
  - BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - BC Cancer Agency - Vancouver Island, Victoria, British Columbia

REFERENCES:
- [Derived] Annala M, Taavitsainen S, Khalaf DJ, Vandekerkhove G, Beja K, Sipola J, Warner EW, Herberts C, Wong A, Fu S, Finch DL, Oja CD, Vergidis J, Zulfiqar M, Eigl BJ, Kollmansberger CK, Nykter M, Gleave ME, Chi KN, Wyatt AW. Evolution of Castration-Resistant Prostate Cancer in ctDNA during Sequential Androgen Receptor Pathway Inhibition. Clin Cancer Res. 2021 Aug 15;27(16):4610-4623. doi: 10.1158/1078-0432.CCR-21-1625. Epub 2021 Jun 3. PMID 34083234
- [Derived] Jayaram A, Wingate A, Wetterskog D, Conteduca V, Khalaf D, Sharabiani MTA, Calabro F, Barwell L, Feyerabend S, Grande E, Martinez-Carrasco A, Font A, Berruti A, Sternberg CN, Jones R, Lefresne F, Lahaye M, Thomas S, Joshi S, Shen D, Ricci D, Gormley M, Merseburger AS, Tombal B, Annala M, Chi KN, De Giorgi U, Gonzalez-Billalabeitia E, Wyatt AW, Attard G. Plasma Androgen Receptor Copy Number Status at Emergence of Metastatic Castration-Resistant Prostate Cancer: A Pooled Multicohort Analysis. JCO Precis Oncol. 2019 Sep 24;3:PO.19.00123. doi: 10.1200/PO.19.00123. eCollection 2019. PMID 32923850
- [Derived] Khalaf DJ, Annala M, Taavitsainen S, Finch DL, Oja C, Vergidis J, Zulfiqar M, Sunderland K, Azad AA, Kollmannsberger CK, Eigl BJ, Noonan K, Wadhwa D, Attwell A, Keith B, Ellard SL, Le L, Gleave ME, Wyatt AW, Chi KN. Optimal sequencing of enzalutamide and abiraterone acetate plus prednisone in metastatic castration-resistant prostate cancer: a multicentre, randomised, open-label, phase 2, crossover trial. Lancet Oncol. 2019 Dec;20(12):1730-1739. doi: 10.1016/S1470-2045(19)30688-6. Epub 2019 Nov 11. PMID 31727538
- [Derived] Khalaf DJ, Sunderland K, Eigl BJ, Kollmannsberger CK, Ivanov N, Finch DL, Oja C, Vergidis J, Zulfiqar M, Gleave ME, Chi KN. Health-related Quality of Life for Abiraterone Plus Prednisone Versus Enzalutamide in Patients with Metastatic Castration-resistant Prostate Cancer: Results from a Phase II Randomized Trial. Eur Urol. 2019 Jun;75(6):940-947. doi: 10.1016/j.eururo.2018.12.015. Epub 2018 Dec 24. PMID 30591354

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT02125357/Prot_SAP_000.pdf